CLINICAL TRIAL: NCT00454883
Title: Treatment Of Manic Or Mixed Episodes Of Up To Moderate Severity In Patients With Bipolar Disorder And Schizoaffective Disorder
Brief Title: Non-interventional Study of Ziprasidone in the Treatment of Bipolar and Schizoaffective Disorders.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281159
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Affective Psychosis, Bipolar; Mania; Manic-Depressive Psychosis
Keywords: Safety of ziprasidone, efficacy of ziprasidone, manic episodes in bipolar disorder, mixed episodes in bipolar disorder, schizoaffective disorder.
MeSH Terms: conditions — Bipolar Disorder; Mania; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 cohort of patients treated with ziprasidone
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Ziprasidone 40 mg twice daily taken with food. Daily dosage may subsequently be adjusted on the basis of individual clinical status up to a maximum of 80 mg twice daily. If indicated, the maximum recommended dose may be reached as early as day 3 of treatment.
  Other Names: Geodon, Zeldox

SUMMARY:
Assessment of ziprasidone safety and efficacy in the treatment of bipolar and schizoaffective disorders.

DETAILED DESCRIPTION:
Method: Consecutive patient sampling. Patients were included in the study in consecutive manner if they fulfilled the inclusion criteria and any of the exclusion criteria were not present.

ELIGIBILITY:
Inclusion Criteria:

* Manic and mixed episodes of up to moderate severity in patients with Type I and II bipolar disorder and schizoaffective disorder; either first diagnosed or repeated episodes

Exclusion Criteria:

* Hypersensitivity to ziprasidone
* prolonged QTc interval
* coadministration with substances that are prolonging the QTc interval
* recent acute MI, cardiac failure, patients with arrhythmias treated with class IA or III medicaments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were identified in in- and outpatients settings (university departments, hospital wards, outpatients clinics, daily psychiatric hospitals)
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Clinical global impression | 3 months
Recording of extrapyramidal symptoms | 3 months
Changes in manic symptoms over course of treatment | 3 months

SECONDARY OUTCOMES:
Severity of disease | 3 months
Adverse Events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281159&StudyName=Non-interventional%20study%20of%20ziprasidone%20in%20the%20treatment%20of%20bipolar%20and%20schizoaffective%20disorders.